CLINICAL TRIAL: NCT04623658
Title: Improving Prenatal Parental Counseling in Cases of Sacrococcygeal Teratoma: a Multicenter Retrospective Study With Review of the Literature
Brief Title: Improving Prenatal Parental Counseling in Cases of Sacrococcygeal Teratoma
Acronym: PROSTEO
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP200355
Record Dates: First submitted 2020-10-28; First posted 2020-11-10 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-09

CONDITIONS: Sacrococcygeal Teratoma
Keywords: Sacrococcygeal teratoma; Prenatal diagnosis; Prenatal counseling; Prognostic factors; Neonatal tumor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sacrococcygeal teratoma: Fetuses and infants diagnosed with sacrococcygeal teratoma and cared for between 2007 and 2017 in the main Parisian fetal medicine and pediatric surgery units: Necker-Enfants Malades Hospital, Antoine Béclère Hospital, Armand Trousseau Hospital, Robert Debré Hospital and Le Kremlin-Bicêtre Hospital.

SUMMARY:
Sacrococcygeal teratoma (SCT) is the most common fetal and neonatal tumor. However, predicting factors of evolution, sequelae and relapse are still unreliable because of small-cohort studies. This study aims at identifying prenatal and postnatal prognostic factors of evolution of SCT during pregnancy, of postnatal relapse, and of medium and long-term sequelae (urinary, digestive, esthetic, psychologic) in order to improve parental counseling when the diagnosis of SCT is made during pregnancy.

DETAILED DESCRIPTION:
Sacrococcygeal teratoma (SCT) is the most common fetal and neonatal tumor. Although mostly benign, SCT can lead to perinatal mortality and long-term sequelae.

Three main risks occur throughout the evolution of SCT:

1. A perinatal life-threatening risk related to the importance of vascularization since SCT can lead to a true arteriovenous fistula with the risk of cardiac failure
2. A risk of benign or malignant tumor recurrence
3. A risk of medium and long-term sequelae, mostly urinary and/or digestive disorders but also aesthetic and psychologic.

In most cases, a prenatal diagnosis is made for which physicians are expected to give a prognosis and counsel parents about medium and long-term complications. However, there is no robust data to date correlating prenatal and postnatal features to prenatal and postnatal evolution of the tumor. The situation is all the more delicate as the information given by the physician can lead to the parent's will to terminate the pregnancy. This retrospective multicentric study aims at identifying prenatal and postnatal prognostic factors of SCT evolution during pregnancy, the occurrence of postnatal relapse after surgical excision, and medium- and long-term sequelae. The primary goal of this study is to improve prenatal parental counseling when the diagnosis of SCT is made.

ELIGIBILITY:
Inclusion Criteria:

* Fetuses and infants (< 1 year) diagnosed with benign sacrococcygeal teratoma
* Cared for between January 2007 and December 2017 in the participating centers

Exclusion Criteria:

* Currarino syndrome
* Other benign sacrococcygeal teratoma discovered after 1 year old or malignant sacrococcygeal tumors

Max Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Fetuses and infants diagnosed with sacrococcygeal teratoma and cared for between 2007 and 2017 in the main Parisian fetal medicine and pediatric surgery units: Necker-Enfants Malades Hospital, Antoine Béclère Hospital, Armand Trousseau Hospital, Robert Debré Hospital and Le Kremlin-Bicêtre Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Presence of postnatal sequelae | Up to 10 years
  Presence of digestive, urinary, cosmetic or psychologic postnatal sequelae
Fetal or neonatal death | Before 28 days of life
  Intrauterine fetal death, termination of pregnancy or neonatal death
Occurrence of benign or malignant recurrence | Up to 10 years
  Relapse requiring subsequent surgical procedures and/or chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Sarnacki, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Nicolas Vinit, Resident, MSc, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Necker-Enfants Malades Hospital, Paris, France

REFERENCES:
- [Result] Vinit N, Bonnard A, Irtan S, Fouquet V, Ville Y, Rosenblatt J, Jouannic JM, Benachi A, Khen-Dunlop N, Lapillonne A, Beaudoin S, Rousseau V, Salomon LJ, Sarnacki S. Perinatal Prognostic Factors of Recurrence or Functional Sequelae in Neonatal Sacrococcygeal Teratoma, and Implications for Prenatal Counselling: A Multicenter Retrospective Study. J Pediatr Surg. 2025 Dec;60(12):162687. doi: 10.1016/j.jpedsurg.2025.162687. Epub 2025 Sep 17. PMID 40972984
- [Result] Vinit N, Benachi A, Rosenblatt J, Jouannic JM, Rousseau V, Bonnard A, Irtan S, Fouquet V, Ville Y, Khen-Dunlop N, Lapillonne A, Jais JP, Beaudoin S, Salomon LJ, Sarnacki S. Growth velocity of fetal sacrococcygeal teratoma as predictor of perinatal morbidity and mortality: multicenter study. Ultrasound Obstet Gynecol. 2024 Nov;64(5):651-660. doi: 10.1002/uog.29110. PMID 39482803